CLINICAL TRIAL: NCT04031053
Title: Assessment of Itraconazole Pharmacokinetic With and Without Efavirenz Using the Capsule Formulation as Part of Talaromycosis Treatment in HIV-infected Adults
Brief Title: Itraconazole Pharmacokinetic With and Without Efavirenz Using the Capsule Formulation as Part of Talaromycosis Treatment in HIV-infected Adults
Acronym: ITRAPK
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chiang Mai University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Quanhathai Kaewpoowat, Principal Investigator, Chiang Mai University
Other Study IDs: ITRAPK
Record Dates: First submitted 2019-04-25; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: Pharmacokinetics; Efavirenz; Penicilliosis
Keywords: Pharmacokinetics; Efavirenz; Penicilliosis
MeSH Terms: conditions — talaromycosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The plasma is stored for drug level analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Pharmacokinetic Group: After receiving the first dose of ITZ, a single blood sample will be collected 12-hours post-dose. On Day 7, the blood will be collected for intensive PK study. After 7 days of combined ITZ + EFV, a blood sample will be collected immediately (e.g. within 30 minutes) prior to administering the next ITZ dose. An identical set of intensive PK blood samples will be drawn 2 weeks after initiating the EFV based regimen.
  Interventions: Other: Pharmacokinetic study
- Trough Level Group: On Days 7 and 14, a single blood sample will be collected immediately (e.g. within 30 minutes) prior to administering the next ITZ dose. After initiating an EFV based regimen, a single blood sample will be collected immediately (e.g. within 30 minutes) prior to administering the next ITZ dose on Days 7 and 14.
  Interventions: Other: Pharmacokinetic study

INTERVENTIONS:
Other: Pharmacokinetic study — The blood will be collected at pre-dose and at 1, 3, 4, 5, 6, 8 and 12-hour post dose

SUMMARY:
Talaromycosis continues to be a common opportunistic fungal infection among people living with HIV/AIDS (PLWHA) in Southeast Asia and remains a leading cause of death among this population. Itraconazole (ITZ) is an important component of talaromycosis treatment. In Thailand, the capsule formulation of ITZ is primarily used to treat talaromycosis but it is known to have lower bioavailability than the more expensive solution formulation. Limited data on the drug exposure of ITZ with the capsule formulation are available in adults PLWHA in Thailand. Moreover, the effect of efavirenz (EFV), which has been recommended as the first line antiretroviral therapy in Thailand, to ITZ level is not well understood. Thus, our aim is to assess ITZ pharmacokinetics with and without EFV in adult PLWHA receiving talaromycosis treatment with the capsule formulation. An understanding of the relationship between ITZ drug exposure and its active metabolite (hydroxyl-itraconazole) and treatment response is also planned to help optimize therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Available documentation of HIV infection
3. ITZ capsule therapy is indicated for talaromycosis infection with the anticipation to start on EFV-based ART
4. Willing to consent and compliance to the study protocol

Exclusion Criteria:

1. History of ITZ allergy
2. Pregnancy or lactation
3. Use concurrent medication that could interfere with ITZ level
4. Creatinine clearance less than 30 mL/min
5. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) value is more than 5 times of upper normal limit and total bilirubin is more than 3 times above upper normal limit
6. Hemoglobin less than 7 mg/dL
7. History of ITZ exposure within 35 days (only applicable to intense PK group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected participant who has an evidence of T. marneffei invasive infection will be enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Itraconazole and its metabolites level | 45 days
  Itraconazole and its metabolite level will be measured to create drug level curve (before and after exposed to efavirenz)

CONTACTS AND LOCATIONS:
Overall Officials: Quanhathai Kaewpoowat, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided